CLINICAL TRIAL: NCT07011290
Title: Physical and Physiological Demands, and Perceived Experience Across Different Recreational Team Handball and Walking Exercise Modalities
Brief Title: Physical and Physiological Demands of Different Recreational Team Handball and Walking Modalitiesmodalities
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Institute of Maia (Other)
Responsible Party: Principal Investigator, Susana Cristina Araújo Póvoas, Associate professor, University Institute of Maia
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 236/2024
Record Dates: First submitted 2025-03-19; First posted 2025-06-08 (Actual); Last update posted 2025-06-08 (Actual); Status verified 2025-05

CONDITIONS: Physiological Demands; Elderly
Keywords: Recreational walking handball; Older adults; Recreational team handball

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Self-paced walking (W) (Other): Each participant will walk at a self-chosen speed during the set exercise duration.
  Interventions: Other: Self-paced Walking (W) training sessions
- Brisk walking (BW) (Other): Participants will walk at a designated speed corresponding to brisk walking ( moderate-intensity walking) during the set exercise duration. The intensity of this type of walking should allow the participants to talk but not sing during the walk.
  Interventions: Other: Brisk walking (BW) training sessions
- Recreational running team handball (RTH) (Other): Participants will play running recreational team handball (RTH) with the following adaptations to the official rules: use of softer and smaller balls and limited body contact, dribbling and substitutions are not allowed; players rotate positions every 3 min and matches are played as 5v5 or 6v6 game formats.
  Interventions: Other: Recreational running team handball (RTH) training sessions
- Recreational walking team handball (WTH) (Other): Same as recreational running team handball (RTH), however, the participants are only permitted to walk and not run (one foot must always be in contact with the ground).
  Interventions: Other: Recreational walking team handball (WTH) training sessions

INTERVENTIONS:
Other: Self-paced Walking (W) training sessions — Participants will partake in 2 sessions of self-paced walking (W), each composed by 3x14 min periods interspersed by 2 min breaks, in which the participants will walk at a self-selected speed (without running) along a 38x18 m course.
  Arms: Self-paced walking (W)
Other: Brisk walking (BW) training sessions — Participants will partake in 2 sessions of brisk walking (BW), each composed by 3x14 min periods, interspersed by 2 min breaks, in which the participants will follow a designated instructor who will dictate the walking speed along a 38x18 m course, thus ensuring that the speed of the walking corresponds to a brisk walking speed.
  Arms: Brisk walking (BW)
Other: Recreational running team handball (RTH) training sessions — Recreational running team handball (RTH):
  Participants will partake in 2 sessions of recreational team handball matches (RTH), each composed by 3x14 min periods, interspersed by 2 min breaks on a 40x20m indoor court.
  Arms: Recreational running team handball (RTH)
Other: Recreational walking team handball (WTH) training sessions — Recreational walking team handball (WTH):
  Participants will partake in 2 sessions of recreational walking team handball matches (WTH), each composed by 3x14 min periods, interspersed by 2 min breaks on a 40x20m indoor court.
  Arms: Recreational walking team handball (WTH)

SUMMARY:
This study aims to determine the physical and physiological demands and perceived experience during different recreational team handball and walking exercise modalities.

Secondary purposes are:

i) To compare the cardiovascular and blood lactate responses to self-paced walking (W), brisk walking (BW), recreational walking team handball (WTH), and recreational running team handball (RTH); ii) To compare the perceived experience (Rating of Perceived Exertion (RPE) and Fun levels (FUN)) during self-paced walking (W), brisk walking (BW), recreational walking team handball (WTH), and recreational running team handball (RTH); iii) To compare the activity profile during self-paced walking (W), brisk walking (BW), recreational walking team handball (WTH), and recreational running team handball (RTH);

DETAILED DESCRIPTION:
Statistical analysis:

Linear mixed-effects model accounting for repeated measures within the participants, will be used to compare the working demands and perceived experience during the selected exercise modalities. This model will consider the exercise modalities and group as fixed effects and the participants ID as a random effect.

Significance level will be set at 5%, and confidence intervals will be reported for all comparisons.

Randomization:

Participants will be randomly assigned to one of two groups due to logistical constraints. Each group will then perform 2 randomly assigned sequences of 4 exercise modalities (i.e., W, BW, WH, RH).

ELIGIBILITY:
Inclusion Criteria:

* Males with 50-82 years
* Previous recreational team handball experience( at least 3 months)

Exclusion Criteria:

* Had any sort of limitation that prevented them from running or gripping a team handball ball
* Had medical contradictions to partake in moderate-to-vigorous physical activity

Ages: 50 Years to 82 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 23 (Estimated)
Dates: Start 2025-03-20 (Actual); Primary Completion 2025-06-17 (Estimated); Study Completion 2025-06-17 (Estimated)

PRIMARY OUTCOMES:
Relative average rate | Over an 8-week period.
  During each exercise modality, relative average rate will be determined using heart rate monitors.
Relative time spent in each heart rate zone | Over an 8-week period.
  During each exercise modality, relative time spent in each heart rate zone will be determined using heart rate monitors.

SECONDARY OUTCOMES:
Absolute average heart rate | Over an 8-week period.
  During each exercise modality, absolute average heart rate will be determined using heart rate monitors.
Absolute time spent in each heart rate zone | Over an 8-week period.
  During each exercise modality, absolute time spent in each heart rate zone will be determined using heart rate monitors.
Relative peak heart rate | Over an 8-week period.
  During each exercise modality, relative peak heart rate will be determined using heart rate monitors.
Absolute peak heart rate | Over an 8-week period.
  During each exercise modality, absolute peak heart rate will be determined using heart rate monitors.
Rating of perceived exertion | Over an 8-week period.
  Rating of perceived exertion (RPE) will be determined using the modified (0-10) Borg scale, during each exercise modality.
Fun levels | Over an 8-week period.
  Fun levels (FUN) will be determined using an visual analog scale, during each exercise modality.
Blood lactate | Over an 8-week period.
  Blood lactate will be measured during the each exercise modality using a portable eletroenzymatic lactate device analyzer.
Accelerations | Over an 8-week period
  The number of accelerations (expressed in m/s²) will be determined during each exercise modality training session using wearable accelerometers. Acceleration thresholds will be defined individually based on activity profiles established in baseline testing.
Decelerations | Over an 8-week period.
  The number of decelerations (expressed in m/s²) will be determined during each exercise modality training session using wearable accelerometers. Deceleration thresholds will be defined individually based on activity profiles established in baseline testing.
Player load | Over an 8-week period.
  Player load (arbitrary units) will be calculated using data from wearable accelerometers during each exercise modality training session.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Maia, Maia, Portugal

IPD SHARING:
Plan to Share IPD: No